CLINICAL TRIAL: NCT01101451
Title: Randomized Phase III Clinical Trial of Adjuvant Radiation Versus Chemoradiation in Intermediate Risk, Stage I/IIA Cervical Cancer Treated With Initial Radical Hysterectomy and Pelvic Lymphadenectomy (NCT #01101451)
Brief Title: Radiation Therapy With or Without Chemotherapy in Patients With Stage I-IIA Cervical Cancer Who Previously Underwent Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0263; NCI-2011-02037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0263 (Other: NRG Oncology); GOG-0263 (Other: CTEP)
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage I Cervical Cancer AJCC v6 and v7; Stage IA Cervical Cancer AJCC v6 and v7; Stage IB Cervical Cancer AJCC v6 and v7; Stage IIA Cervical Cancer AJCC v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiation; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (EBRT, IMRT) (Active Comparator): Patients undergo pelvic EBRT or IMRT once daily, 5 days a week, for 5.5 weeks.
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (cisplatin, EBRT, IMRT) (Experimental): Patients receive cisplatin IV over 1-2 hours on day 1 and undergo radiotherapy as in Arm I. Treatment with cisplatin repeats every 7 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm II (cisplatin, EBRT, IMRT)
Radiation: External Beam Radiation Therapy — Undergo radiotherapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
Radiation: Intensity-Modulated Radiation Therapy — Undergo radiotherapy
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies radiation therapy with chemotherapy to see how well they work compared to radiation therapy alone in treating patients with stage I-IIA cervical cancer who previously underwent surgery. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving radiation therapy together with chemotherapy is more effective than radiation therapy alone in treating patients with cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if post-operative adjuvant chemo-radiation therapy (CRT) can significantly improve recurrence-free survival (RFS) when compared to radiation therapy (RT) alone in stage I-IIA cervical cancer patients with intermediate-risk factors after treatment with radical hysterectomy.

SECONDARY OBJECTIVES:

I. To determine whether post-operative adjuvant CRT can improve overall survival (OS) when compared to RT alone in stage I-IIA cervical cancer patients with intermediate risk factors after treatment with radical hysterectomy.

II. To assess differences (across treatment arms) in incidence and severity of therapy attributed adverse events utilizing the active version of Common Terminology Criteria for Adverse Events (CTCAE).

III. To provide assessment of patient risk version (vs) benefit (positive study only).

QUALITY OF LIFE OBJECTIVE:

I. To determine whether post-operative adjuvant CRT improves the health-related quality-of-life (QOL) (compared to RT alone) as measured by Functional Assessment of Cancer Therapy-Cervix (FACT-Cx) Trial Outcome Index (TOI) and produce favorable toxicity profiles (with particular focus on treatment related genitourinary, gastrointestinal, neurological, pain and sexual adverse events).

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To bank archival tumor tissue for research studies, including studies that evaluate the association between biomarkers, RFS, OS, and clinical-surgical-pathologic characteristics in patients randomized to post-operative adjuvant CRT compared to RT alone.

II. To bank deoxyribonucleic acid (DNA) from whole blood for research studies, including studies that evaluate associations between single nucleotide polymorphisms (SNPs), and measures of clinical outcome, including RFS, OS, and adverse events in patients randomized to post-operative adjuvant CRT compared to RT alone.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo pelvic external-beam radiation therapy (EBRT) or intensity-modulated radiation therapy (IMRT) 5 days a week for 5.5 weeks.

ARM II: Patients receive cisplatin IV over 1-2 hours on day 1 and undergo radiotherapy as in Arm I. Treatment with cisplatin repeats every 7 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven primary cervical cancer I-IIA with squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma initially treated with a standard radical hysterectomy with pelvic lymphadenectomy
* Patients with the following characteristics (depth of stromal invasion and lymphovascular space involvement to be pathologically confirmed):

  * Positive capillary-lymphovascular space involvement and one of the following:

    * Deep third penetration
    * Middle third penetration, clinical tumor >= 2 cm
    * Superficial third penetration, clinical tumor >= 5 cm
  * Negative capillary-lymphatic space involvement

    * Middle or deep third penetration, clinical tumor >= 4 cm
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 100,000/mcl
* Creatinine =< upper limit of normal (ULN) or calculated creatinine clearance >= 60 mL/min
* Bilirubin =< 1.5 x normal
* Alkaline phosphate =< 3 x normal
* Serum glutamic oxaloacetic transaminase (SGOT) =< 3 x normal
* Gynecologic Oncology Group (GOG) performance status 0, 1, 2
* Patients should not be randomized less than 3 weeks post-surgery but will not be acceptable for randomization more than 8 weeks post-surgery
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with tumor in the parametria, pelvic lymph nodes or any other extra uterine site or with positive surgical margins
* Patients with septicemia or severe infection
* Patients with intestinal obstruction or gastrointestinal bleeding
* Patients with postoperative fistula
* Patients with cervix cancer who have received any previous radiation or chemotherapy
* Patients whose circumstances do not permit completion of the study or the required follow-up
* Patients with renal abnormalities requiring modification of radiation field (pelvic kidney, renal transplant, etc.)
* Patients with GOG performance status of 3 or 4
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2010-04-12 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Y Ryu, Principal Investigator — NRG Oncology
Locations (719):
- United States (698):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Sutter Davis Hospital, Davis, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Abben Cancer Center, Spencer, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Austin Cancer Centers-Central Austin, Austin, Texas
  - Austin Cancer Centers-North, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Japan (8):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure National Hospital, Kure, Hiroshima
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Shizuoka Cancer Center, Shizuoka, Suntou
  - Shikoku Cancer Center, Matsuyama
  - Kindai University, Osaka
- South Korea (13):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Inha University, Jung-gu, Incheon
  - Samsung Medical Center, Seoul, Korea
  - Catholic University of Korea-Seoul Saint Mary's Hospital, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System-Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Korea Cancer Center Hospital, Seoul

REFERENCES:
- [Derived] Kim H, Park W, Kim YS, Kim YJ. Chemoradiotherapy is not superior to radiotherapy alone after radical surgery for cervical cancer patients with intermediate-risk factor. J Gynecol Oncol. 2020 May;31(3):e35. doi: 10.3802/jgo.2020.31.e35. Epub 2019 Nov 21. PMID 31912685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG-0263 opened to accrual on April 12, 2010, and closed to accrual on April 11, 2022.
Groups:
- Arm I (Radiation): Patients undergo pelvic external-beam radiation therapy (EBRT) or intensity-modulated radiation therapy (IMRT) 5 days a week for 5.5 weeks.
- Arm II (Cisplatin + Radiation): Patients receive cisplatin IV over 1-2 hours on day 1 and undergo radiotherapy as in Arm I. Treatment with cisplatin repeats every 7 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
Started | 172 | 168
Completed | 158 | 153
Not Completed | 14 | 15
Not completed — Eligible and never treated | 0 | 5
Not completed — Ineligible and treated | 12 | 8
Not completed — Ineligible and never treated | 2 | 2

BASELINE CHARACTERISTICS:
Population: Eligible
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation) | Total
Number analyzed (Participants) | 158 | 158 | 316
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 3 | 2 | 5
  30-39 years | 28 | 47 | 75
  40-49 years | 62 | 53 | 115
  50-59 years | 46 | 33 | 79
  60-69 years | 13 | 17 | 30
  70-79 years | 5 | 6 | 11
  >= 80 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 158 | 316
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 142 | 142 | 284
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 79 | 87 | 166
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 5 | 17
  White | 62 | 58 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS) Rate at 3-years
Description: Estimate for probability of RFS at 3 years using Kaplan-Meier method, where RFS is defined as time from protocol registration (and randomization) to the date of first documented recurrence, death, or the date of last contact, whichever occurs first. Patients without recurrence or death were censored at the date of last contact.
Time Frame: 3 years from randomization
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
Number analyzed (Participants) | 158 | 158
percentage of participants | 85.4 [79 to 90] | 88.5 [82 to 93]
Statistical Analysis 1: Comparison: Arm I (Radiation) vs Arm II (Cisplatin + Radiation); Test type: Superiority; p = 0.0927, Log Rank — the pre_specified nominal significance level was 0.0451 (one sided); Hazard Ratio (HR) = 0.6976, 95% CI 2-sided [0.408 to 1.192] — The RFS hazard ratio estimate is for reporting group 2 vs reporting group 1

2. Secondary Outcome: Overall Survival (OS) Rate at 3-years
Description: Estimate for probability of overall survival at 3 years by Kaplan-Meier method, where overall survival is defined as the time from randomization to time of death due to any cause or the date of last contact, whichever occurs first.
Time Frame: 3 years from randomization
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
Number analyzed (Participants) | 158 | 158
percentage of participants | 90.3 [84 to 94] | 97.2 [93 to 99]
Statistical Analysis 1: Comparison: Arm I (Radiation) vs Arm II (Cisplatin + Radiation); Test type: Superiority; Hazard Ratio (HR) = 0.586, 95% CI 2-sided [0.286 to 1.199] — The OS hazard ratio estimate is for reporting group 2 vs reporting group 1

3. Secondary Outcome: Number of Participants With Adverse Events (Grade 3 or Higher) During Treatment Period.
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: During treatment period and up to 21 days after stopping the study treatment. The median treatment duration was 39 days.
Population: Randomized participants who received any assigned protocol therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
Number analyzed (Participants) | 170 | 161
Participants
  Anemia | 1 | 6
  Other blood/lymphatics | 0 | 4
  White blood cell decreased | 3 | 45
  Platelet count decreased | 0 | 4
  Neutrophil count decreased | 2 | 27
  Other investigations | 7 | 8
  Gastrointestinal | 10 | 12
  General and administration site | 2 | 3
  Infections/infestations | 4 | 4
  Metabolism/nutrition | 0 | 7
  Musculoskeletal/connective tissue | 1 | 0
  Nervous system | 2 | 1
  Psychiatric | 1 | 1
  Renal/urinary | 2 | 2
  Reproductive/breast | 2 | 1
  Skin/subcutaneous | 0 | 3
  Vascular disorders | 0 | 1

4. Secondary Outcome: Patient Risk-benefit
Description: The reporting group (2) did not demonstrate improved RFS compared to the reporting group (1) at the pre-specified significance level. Per the protocol, patient risk-benefit will be assessed only for a positive study.
  This is not assessed due to non-positive study per the protocol.
Time Frame: up to 11 years
Population: Per protocol, patient risk-benefit will be assessed only for a positive study. Based on the results information at the specified significance level, patient risk-benefit was not assessed as pre-specified
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life (QOL) as Measured With the FACT-Cx TOI
Description: The patient-reported QOL is assessed with the Trial Outcome Index of the Functional Assessment of Cancer Therapy-Cervix (FACT-Cx TOI). The FACT-Cx TOI is ranged 0-116 and a larger FACT-Cx TOI score suggests a favorable QoL.
Time Frame: 1. Pre-treatment (baseline), 2. 3 weeks following the first day of treatment, 3. 7 weeks following the first day of treatment, 4. 36 weeks following the first day of treatment.
Population: Eligible patients who completed baseline and at lease one follow-up QOL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
Number analyzed (Participants) | 152 | 147
units on a scale
  Baseline | 83.5 (15.4) | 80.1 (15.4)
  3 weeks | 79.0 (16.4) | 71.4 (15.3)
  7 weeks | 80.1 (17.0) | 71.8 (17.1)
  36 weeks | 88.8 (15.5) | 88.1 (12.3)

6. Other Pre Specified Outcome: Treatment Compliance
Description: Assessed by the number of cycles and amount of chemoradiotherapy administered, treatment span, incidence and duration of treatment delays, reason for delays, and reason why off study therapy.
Time Frame: Up to 11 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Site(s) of Recurrence
Description: The site(s) of first disease recurrence will be classified as: pelvic-only, extra-pelvic-only or pelvic-and-extra-pelvic and tabulated by treatment group. The test of the hypothesis that the probability of local failure is independent of randomized treatment will be assessed with exact logistic regression adjusted know prognostic factors.
Time Frame: Up to 11 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Local Control
Description: Assessed with Exact Logistic Regression adjusted known prognostic factors.
Time Frame: Up to 11 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During treatment period and up to 21 days after stopping the study treatment. The median treatment duration was 39 days.
Description: All randomized participants who received any assigned protocol therapy were monitored/assessed for serious adverse events and other adverse events. Randomized eligible participants were monitored/assessed for All-Cause Mortality.
  The All-Cause Mortality that occurred from randomization until 54 RFS events have occurred with a median follow-up 76.5 months (inter-quartile range: 50.3 to 107.7 months) estimated by reverse Kaplan-Meier method.
Arm/Group | Arm I (Radiation) | Arm II (Cisplatin + Radiation)
All-Cause Mortality (participants affected / at risk) | 20/158 | 12/158
Serious Adverse Events (participants affected / at risk) | 7/170 | 9/161
Other Adverse Events (participants affected / at risk) | 140/170 | 158/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Radiation) (N=170) | Arm II (Cisplatin + Radiation) (N=161)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Colonic Fistula (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Infections And Infestations - Other (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
White Blood Cell Decreased (Investigations) | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 1
Vaginal Pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Radiation) (N=170) | Arm II (Cisplatin + Radiation) (N=161)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 | 5
Anemia (Blood and lymphatic system disorders) | 63 | 95
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 5
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 | 0
Chest Pain - Cardiac (Cardiac disorders) | 0 | 1
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 19
Ear Pain (Ear and labyrinth disorders) | 0 | 3
Endocrine Disorders - Other (Endocrine disorders) | 0 | 1
Eye Disorders - Other (Eye disorders) | 1 | 1
Flashing Lights (Eye disorders) | 0 | 2
Eye Pain (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 0 | 6
Floaters (Eye disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 11
Constipation (Gastrointestinal disorders) | 26 | 63
Diarrhea (Gastrointestinal disorders) | 76 | 78
Vomiting (Gastrointestinal disorders) | 14 | 37
Bloating (Gastrointestinal disorders) | 0 | 2
Stomach Pain (Gastrointestinal disorders) | 1 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 28 | 23
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Mucositis Oral (Gastrointestinal disorders) | 0 | 2
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 2 | 0
Anal Pain (Gastrointestinal disorders) | 17 | 12
Oral Pain (Gastrointestinal disorders) | 0 | 3
Abdominal Distension (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 61 | 117
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 5
Rectal Pain (Gastrointestinal disorders) | 3 | 3
Fecal Incontinence (Gastrointestinal disorders) | 2 | 1
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 8 | 10
Malaise (General disorders) | 3 | 7
Localized Edema (General disorders) | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 4 | 5
Edema Trunk (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Edema Limbs (General disorders) | 10 | 5
Edema Face (General disorders) | 1 | 0
Fatigue (General disorders) | 46 | 74
Fever (General disorders) | 2 | 14
Chills (General disorders) | 0 | 4
Infusion Related Reaction (General disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 0 | 3
Immune System Disorders - Other (Immune system disorders) | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 0 | 2
Upper Respiratory Infection (Infections and infestations) | 1 | 1
Vulval Infection (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 1 | 1
Lymph Gland Infection (Infections and infestations) | 1 | 0
Pelvic Infection (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Vaginal Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 12 | 14
Bladder Infection (Infections and infestations) | 1 | 5
Anorectal Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis Radiation (Injury, poisoning and procedural complications) | 2 | 5
Bruising (Injury, poisoning and procedural complications) | 0 | 3
Investigations - Other (Investigations) | 0 | 4
Weight Loss (Investigations) | 3 | 4
Weight Gain (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 19 | 73
Lymphocyte Count Decreased (Investigations) | 9 | 10
Creatinine Increased (Investigations) | 0 | 7
Neutrophil Count Decreased (Investigations) | 36 | 88
Blood Bilirubin Increased (Investigations) | 1 | 0
White Blood Cell Decreased (Investigations) | 73 | 121
Aspartate Aminotransferase Increased (Investigations) | 0 | 4
Alkaline Phosphatase Increased (Investigations) | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 8
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 11
Hypokalemia (Metabolism and nutrition disorders) | 4 | 14
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 18 | 48
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous System Disorders - Other (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 | 13
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 2
Meningismus (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 27
Dysgeusia (Nervous system disorders) | 3 | 13
Sinus Pain (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 16
Acoustic Nerve Disorder Nos (Nervous system disorders) | 0 | 1
Psychiatric Disorders - Other (Psychiatric disorders) | 1 | 1
Personality Change (Psychiatric disorders) | 1 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 19
Depression (Psychiatric disorders) | 2 | 7
Anxiety (Psychiatric disorders) | 5 | 10
Agitation (Psychiatric disorders) | 2 | 3
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 1 | 3
Urinary Urgency (Renal and urinary disorders) | 5 | 3
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 8 | 6
Urinary Incontinence (Renal and urinary disorders) | 1 | 7
Urinary Tract Pain (Renal and urinary disorders) | 15 | 16
Urinary Frequency (Renal and urinary disorders) | 17 | 18
Proteinuria (Renal and urinary disorders) | 2 | 1
Hematuria (Renal and urinary disorders) | 2 | 2
Cystitis Noninfective (Renal and urinary disorders) | 8 | 13
Bladder Spasm (Renal and urinary disorders) | 2 | 3
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 0 | 1
Vaginal Stricture (Reproductive system and breast disorders) | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 3 | 5
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 3
Vaginal Dryness (Reproductive system and breast disorders) | 2 | 1
Uterine Pain (Reproductive system and breast disorders) | 1 | 0
Perineal Pain (Reproductive system and breast disorders) | 0 | 5
Pelvic Pain (Reproductive system and breast disorders) | 9 | 6
Vaginal Discharge (Reproductive system and breast disorders) | 4 | 6
Dyspareunia (Reproductive system and breast disorders) | 1 | 2
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 3
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Induration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 6
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 9
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1 | 0
Lymphocele (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 5
Hot Flashes (Vascular disorders) | 10 | 12
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT01101451/Prot_SAP_000.pdf